CLINICAL TRIAL: NCT03180684
Title: A Phase 2, Randomized, Open Label, Efficacy Study of VGX-3100 Delivered Intramuscularly Followed by Electroporation With CELLECTRA™ 2000 Alone or in Combination With Imiquimod, for the Treatment of HPV-16 and/or HPV-18 Related High Grade Squamous Intraepithelial Lesion (HSIL) of the Vulva
Brief Title: Evaluation of VGX-3100 and Electroporation Alone or in Combination With Imiquimod for the Treatment of HPV-16 and/or HPV-18 Related Vulvar HSIL (Also Referred as: VIN 2 or VIN 3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPV-201
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Vulvar High Grade Squamous Intraepithelial Lesion (HSIL); Vulvar Dysplasia; Vulvar Intraepithelial Neoplasia (VIN); VIN2; VIN3; Pre-cancerous Lesions of the Vulva; Human Papillomavirus (HPV)
Keywords: HPV-16; HPV-18
MeSH Terms: interventions — VGX-3100; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- VGX-3100 + EP (Experimental): Participants with histologically confirmed vulvar high-grade squamous intraepithelial lesion (HSIL) associated with human papilloma virus (HPV) 16 and/or 18, received four doses of 6 mg VGX-3100 as an intramuscular (IM) injection on Day 0, Week 4, Week 12, and Week 24 followed by electroporation (EP) using the CELLECTRA™ 2000 device. Participants with vulvar HSIL who had a reduction in lesion size or no increase in lesion size at Week 48, received a fifth dose of VGX-3100 at Week 52.
  Interventions: Biological: VGX-3100; Device: CELLECTRA™ 2000
- VGX-3100 + EP + Imiquimod (Experimental): Participants with histologically confirmed vulvar HSIL associated with HPV-16 and/or 18, received four doses of 6 mg VGX-3100 as an IM injection on Day 0, Week 4, Week 12, and Week 24 followed by EP using the CELLECTRA™ 2000 device. Participants with vulvar HSIL who had a reduction in lesion size or no increase in lesion size at Week 48, received a fifth dose of VGX-3100 at Week 52. In addition, participants applied imiquimod 5% cream to the vulvar lesion three times per week for 20 weeks.
  Interventions: Biological: VGX-3100; Drug: Imiquimod 5% Cream; Device: CELLECTRA™ 2000

INTERVENTIONS:
Biological: VGX-3100 — One milliliter (1 mL) VGX-3100 injected IM and delivered by EP using CELLECTRA™ 2000 on Day 0, Week 4, Week 12 and Week 24.
Drug: Imiquimod 5% Cream — Participants applied imiquimod 5% cream to the vulvar lesion three times per week for 20 weeks.
  Arms: VGX-3100 + EP + Imiquimod
Device: CELLECTRA™ 2000 — IM injection of VGX-3100 was followed by EP with the CELLECTRA™ 2000 device.

SUMMARY:
The purpose of this study is to test the safety and efficacy of an investigational immunotherapy VGX-3100, in combination with a study device, to treat women with vulvar high-grade squamous intraepithelial lesion (HSIL) [vulval intraepithelial neoplasia 2 or 3 (VIN 2 or VIN 3)] associated with human papilloma virus (HPV) types 16 and/or 18. VGX-3100 is being assessed as an alternative to surgery with the potential to clear the underlying HPV infection. For more information visit our study website at: www.VINresearchstudy.com

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and above;
* Have high grade squamous intraepithelial lesion (HSIL) of the vulva (VIN2 or VIN3) caused by infection with HPV types 16 and/or 18 confirmed at screening visit;

Exclusion Criteria:

* Biopsy-proven differentiated VIN;
* Any previous treatment for vulvar HSIL within 4 weeks prior to screening;
* Allergy to imiquimod 5% cream or to an inactive ingredient in imiquimod 5% cream;
* Pregnant, breastfeeding or considering becoming pregnant within 6 months following the last dose of investigational product;
* Immunosuppression as a result of underlying illness or treatment;
* Significant acute or chronic medical illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (15):
- United States (15):
  - Christiana Care Health Systems, Newark, Delaware
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Maine Medical Center, Scarborough, Maine
  - University of Michigan, Ann Arbor, Michigan
  - St. Dominic Hospital, Jackson, Mississippi
  - Rutgers New Jersey, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Complete HealthCare for Women, Inc., Columbus, Ohio
  - University of Pittsburgh Medical Center - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 20 study sites in the United States from 31 August 2017 to 18 December 2020.
Pre-assignment Details: A total of 70 participants were screened out of which 33 participants were enrolled in the study.
Period: Overall Study
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Started | 25 | 8
Modified Intent-to-Treat (mITT) Population (mITT population included all participants who received at least 1 dose of VGX-3100 + EP (with or without imiquimod) and had an analysis endpoint of interest.) | 25 | 8
Safety Population (Safety population included all participants who received at least 1 dose of VGX-3100 (with or without EP).) | 25 | 8
Completed | 17 | 8
Not Completed | 8 | 0
Not completed — Withdrawal by Subject (Not Related to AE) | 5 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive Disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: mITT population included all participants who received at least 1 dose of VGX-3100 + EP (with or without imiquimod) and had an analysis endpoint of interest.
Groups:
- VGX-3100 + EP: Participants with histologically confirmed vulvar HSIL associated with HPV-16 and/or 18, received four doses of 6 mg VGX-3100 as an IM injection on Day 0, Week 4, Week 12, and Week 24 followed by EP using the CELLECTRA™ 2000 device. Participants with vulvar HSIL who had a reduction in lesion size or no increase in lesion size at Week 48, received a fifth dose of VGX-3100 at Week 52.
- Total: Total of all reporting groups
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod | Total
Number analyzed (Participants) | 25 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (12.86) | 45.4 (9.13) | 49.1 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 8 | 33
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African | 3 | 0 | 3
  Race: White | 21 | 8 | 29
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Histologic Evidence of Vulvar HSIL and No Evidence of HPV-16 and/or HPV-18 in Vulvar Tissue Samples
Description: A treatment responder for the primary endpoint was defined as a participant with no histologic evidence of vulvar HSIL (normal tissue or vulvar low grade squamous intraepithelial lesions (LSIL) [vulval intraepithelial neoplasia 1 (VIN1)] or condyloma) and no evidence of HPV-16 or HPV-18 (i.e., elimination of the specific genotypes [16, 18, or both]) in vulvar tissue at evaluation and who did not receive any non-study related treatment for vulvar HSIL. All lesions were evaluated for histologic evidence of vulvar HSIL or evidence of HPV-16/18 in vulvar tissue.
Time Frame: Week 48
Population: mITT population included all participants who received at least 1 dose of VGX-3100 + EP (with or without imiquimod) and had an analysis endpoint of interest. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 20 | 8
percentage of participants | 15.0 [3.2 to 37.9] | 37.5 [8.5 to 75.5]
Statistical Analysis 1: Comparison: VGX-3100 + EP; Test type: Superiority; p = 0.0071, Clopper Pearson; A 1-sided p-value was calculated to prove superiority over historical control of 2%. Superiority of VGX-3100 alone was declared if p-value is <0.025
Statistical Analysis 2: Comparison: VGX-3100 + EP + Imiquimod; Test type: Superiority; p = 0.0004, Clopper Pearson; 1-sided p-value was calculated to prove superiority over historical control of 2%.Superiority of VGX-3100+imiquimod was declared if p-value is <0.025

2. Secondary Outcome: Percentage of Participants With at Least One Local and Systemic Treatment-emergent Adverse Event (TEAE) During 7 Days Following Each Dose
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, or worsening of a pre-existing condition, temporally associated with the use of a product whether or not considered related to the use of the product. A TEAE was defined per protocol as any AE with onset after the administration of study medication through the end of the study (i.e., study discharge).
Time Frame: 7 days following each dose: Day 0 (Days 0 to 7), Week 4 (Days 22 to 28), Week 12 (Days 78 to 84), Week 24 (Days 162 to 168), and Week 52 (Days 358 to 364)
Population: Safety population included all participants who received at least one (1) dose of VGX-3100 (with or without EP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 25 | 8
percentage of participants | 84.0 [63.92 to 95.46] | 75.0 [34.91 to 96.81]

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, or worsening of a pre-existing condition, temporally associated with the use of a product whether or not considered related to the use of the product.
Time Frame: From baseline up to Week 100
Population: Safety population included all participants who received at least 1 dose of VGX-3100 (with or without EP).
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 25 | 8
percentage of participants | 92.0 | 100

4. Secondary Outcome: Percentage of Participants With No Histologic Evidence of Vulvar HSIL
Description: Participants with no histologic evidence of vulvar HSIL (normal tissue or vulvar LSIL [VIN1] or condyloma) based on histology (i.e. biopsies or excisional treatment) were considered. All lesions were evaluated for histologic evidence of vulvar HSIL.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 20 | 8
percentage of participants | 15.0 [3.2 to 37.9] | 37.5 [8.5 to 75.5]

5. Secondary Outcome: Percentage of Participants With No Evidence of HPV-16 and/or HPV-18 in Vulvar Tissue Samples
Description: Participants with no evidence of HPV-16 and/or HPV-18 indicated the clearance of the specific HPV genotypes [16, 18, or both]. All lesions were evaluated for evidence of HPV-16/18 in vulvar tissue.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- VGX-3100 + EP + Imiquimod: Participants with histologically confirmed vulvar HSIL associated with HPV-16 and/or 18, received four doses of 6 mg VGX-3100 as an IM injection on Day 0, Week 4, Week 12, and Week 24 followed by EP using the CELLECTRA™ 2000 device. Participants with vulvar HSIL who had a reduction in lesion size or no increase in lesion size at Week 48, received a fifth dose of VGX-3100 at Week 52.
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 20 | 8
percentage of participants | 15.0 [3.2 to 37.9] | 50.0 [15.7 to 84.3]

6. Secondary Outcome: Percentage of Participants With No Histologic Evidence of Vulvar HSIL or No Evidence of HPV-16/18 in Vulvar Tissue
Description: A treatment responder for the endpoint was defined as a participant with no histologic evidence of vulvar HSIL (normal tissue or LSIL [VIN1] or condyloma) based on histology (i.e. biopsies or excisional treatment) or no evidence of HPV-16 or HPV-18 (i.e., elimination of the specific genotypes [16, 18, or both]) in vulvar tissue at evaluation and who did not receive any non-study related treatment for vulvar HSIL. All lesions were evaluated for histologic evidence of vulvar HSIL or evidence of HPV-16/18 in vulvar tissue.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 20 | 8
percentage of participants | 15.0 [3.2 to 37.9] | 50.0 [15.7 to 84.3]

7. Secondary Outcome: Percentage of Participants With No Evidence of Vulvar HSIL, No Evidence of Vulvar LSIL (VIN1), and No Evidence of Condyloma on Histology
Description: Histologic regression was defined as a participant with no histologic evidence of vulvar HSIL, no evidence of LSIL (VIN1), and no evidence of condyloma. Histologic regression of vulvar HSIL to normal tissue was assessed.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 20 | 8
percentage of participants | 10.0 [1.2 to 31.7] | 37.5 [8.5 to 75.5]

8. Secondary Outcome: Percentage of Participants With No Progression of Vulvar HSIL to Vulvar Cancer
Description: Non-progression of vulvar HSIL to vulvar cancer was evaluated from baseline to Week 48. Progression was defined as advancement to carcinoma by histology.
Time Frame: From baseline up to Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 20 | 8
percentage of participants | 100.0 [83.2 to 100.0] | 100.0 [63.1 to 100.0]

9. Secondary Outcome: Percent Change From Baseline in the Cumulative Surface Area of the Acetowhite Vulvar Lesion(s)
Description: Lesion(s), defined as areas that stain acetowhite were assessed. Analysis of qualifying lesions was defined as the change in total surface area of only lesions with both baseline and Week 48 measurements. Percent change in the cumulative surface area of the acetowhite vulvar lesion(s) was determined by the quantitative analysis of standardized prebiopsy photographic imaging of qualifying lesion(s) at Week 48 compared to baseline.
Time Frame: From baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in surface area
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 19 | 7
percent change in surface area | 47.7 (249.62) | 10.5 (117.95)

10. Secondary Outcome: Change From Baseline in Interferon-Gamma (IFN-γ) Response Magnitude
Description: Peripheral blood mononuclear cells (PBMCs) were isolated from whole blood samples. Assessment of cellular immune activity was performed by IFN-γ enzyme-linked immunosorbent spot-forming (ELISpot) assay.
Time Frame: Baseline; Weeks 15, 27, 48, 74, and 96
Population: mITT population included all participants who received at least 1 dose of VGX-3100 + EP (with or without imiquimod) and had an analysis endpoint of interest. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants available for analysis at individual time points.
Measure: Median (Full Range); unit: spot forming units (SFU) per 10^6 cells
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 24 | 7
spot forming units (SFU) per 10^6 cells
  HPV-16 E6 (Baseline) | 1.667 [0.00 to 35.00] | 1.667 [0.00 to 8.33]
  HPV-16 E6 (Change From Baseline at Week 15): number analyzed (Participants) | 22 | 7
  HPV-16 E6 (Change From Baseline at Week 15) | 0.833 [0.00 to 78.33] | 0.000 [0.00 to 43.33]
  HPV-16 E6 (Change From Baseline at Week 27): number analyzed (Participants) | 22 | 7
  HPV-16 E6 (Change From Baseline at Week 27) | 0.833 [0.00 to 58.33] | 3.333 [0.00 to 36.67]
  HPV-16 E6 (Change From Baseline at Week 48): number analyzed (Participants) | 20 | 7
  HPV-16 E6 (Change From Baseline at Week 48) | 0.833 [0.00 to 56.67] | 0.000 [0.00 to 3.33]
  HPV-16 E6 (Change From Baseline at Week 74): number analyzed (Participants) | 15 | 4
  HPV-16 E6 (Change From Baseline at Week 74) | 1.667 [0.00 to 30.00] | 0.000 [0.00 to 25.00]
  HPV-16 E6 (Change From Baseline at Week 96): number analyzed (Participants) | 3 | 4
  HPV-16 E6 (Change From Baseline at Week 96) | 1.667 [0.00 to 38.33] | 0.833 [0.00 to 8.33]
  HPV-16 E7 (Baseline) | 1.667 [0.00 to 15.00] | 0.000 [0.00 to 1.67]
  HPV-16 E7 (Change From Baseline at Week 15): number analyzed (Participants) | 22 | 7
  HPV-16 E7 (Change From Baseline at Week 15) | 3.333 [0.00 to 43.33] | 1.667 [0.00 to 56.67]
  HPV-16 E7 (Change From Baseline at Week 27): number analyzed (Participants) | 22 | 7
  HPV-16 E7 (Change From Baseline at Week 27) | 3.333 [0.00 to 71.67] | 6.667 [0.00 to 40.00]
  HPV-16 E7 (Change From Baseline at Week 48): number analyzed (Participants) | 20 | 7
  HPV-16 E7 (Change From Baseline at Week 48) | 1.667 [0.00 to 31.67] | 1.667 [0.00 to 25.00]
  HPV-16 E7 (Change From Baseline at Week 74): number analyzed (Participants) | 15 | 4
  HPV-16 E7 (Change From Baseline at Week 74) | 1.667 [0.000 to 15.00] | 0.833 [0.00 to 21.67]
  HPV-16 E7 (Change From Baseline at Week 96): number analyzed (Participants) | 3 | 4
  HPV-16 E7 (Change From Baseline at Week 96) | 0.000 [0.000 to 3.33] | 0.000 [0.00 to 0.00]
  HPV-18 E6 (Baseline) | 0.000 [0.00 to 6.67] | 0.000 [0.00 to 6.67]
  HPV-18 E6 (Change From Baseline at Week 15): number analyzed (Participants) | 22 | 7
  HPV-18 E6 (Change From Baseline at Week 15) | 19.167 [0.00 to 593.33] | 10.000 [1.67 to 123.33]
  HPV-18 E6 (Change From Baseline at Week 27): number analyzed (Participants) | 22 | 7
  HPV-18 E6 (Change From Baseline at Week 27) | 10.833 [0.00 to 908.33] | 5.000 [0.00 to 146.67]
  HPV-18 E6 (Change From Baseline at Week 48): number analyzed (Participants) | 20 | 7
  HPV-18 E6 (Change From Baseline at Week 48) | 14.167 [0.00 to 566.67] | 3.333 [0.00 to 80.00]
  HPV-18 E6 (Change From Baseline at Week 74): number analyzed (Participants) | 15 | 4
  HPV-18 E6 (Change From Baseline at Week 74) | 8.333 [0.00 to 925.00] | 9.167 [0.00 to 45.00]
  HPV-18 E6 (Change From Baseline at Week 96): number analyzed (Participants) | 3 | 4
  HPV-18 E6 (Change From Baseline at Week 96) | 20.000 [0.00 to 63.33] | 19.167 [1.67 to 48.33]
  HPV-18 E7 (Baseline) | 0.000 [0.00 to 11.67] | 0.000 [0.00 to 3.33]
  HPV-18 E7 (Change From Baseline at Week 15): number analyzed (Participants) | 22 | 7
  HPV-18 E7 (Change From Baseline at Week 15) | 2.500 [0.00 to 51.67] | 3.333 [0.00 to 16.67]
  HPV-18 E7 (Change From Baseline at Week 27): number analyzed (Participants) | 22 | 7
  HPV-18 E7 (Change From Baseline at Week 27) | 1.667 [0.00 to 33.33] | 6.667 [0.00 to 43.33]
  HPV-18 E7 (Change From Baseline at Week 48): number analyzed (Participants) | 20 | 7
  HPV-18 E7 (Change From Baseline at Week 48) | 1.667 [0.00 to 51.67] | 0.000 [0.00 to 21.67]
  HPV-18 E7 (Change From Baseline at Week 74): number analyzed (Participants) | 15 | 4
  HPV-18 E7 (Change From Baseline at Week 74) | 1.667 [0.00 to 20.00] | 0.000 [0.00 to 6.67]
  HPV-18 E7 (Change From Baseline at Week 96): number analyzed (Participants) | 3 | 4
  HPV-18 E7 (Change From Baseline at Week 96) | 3.333 [0.00 to 5.00] | 4.167 [0.00 to 13.33]

11. Secondary Outcome: Levels of Serum Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations
Description: A standardized binding enzyme-linked immunosorbent assay (ELISA) was performed to measure the anti-HPV-16/18 antibody response induced by VGX-3100.
Time Frame: Weeks 15, 27, 48, 74, and 96
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: reciprocal endpoint titer
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 24 | 8
reciprocal endpoint titer
  Anti-HPV-16 (Week 15): number analyzed (Participants) | 23 | 8
  Anti-HPV-16 (Week 15) | 7.3 (3.22) | 13.1 (2.89)
  Anti-HPV-16 (Week 27) | 9.6 (3.24) | 15.0 (3.07)
  Anti-HPV-16 (Week 48): number analyzed (Participants) | 20 | 8
  Anti-HPV-16 (Week 48) | 15.9 (3.33) | 17.2 (3.06)
  Anti-HPV-16 (Week 74): number analyzed (Participants) | 15 | 6
  Anti-HPV-16 (Week 74) | 14.5 (3.31) | 6.1 (2.80)
  Anti-HPV-16 (Week 96): number analyzed (Participants) | 3 | 4
  Anti-HPV-16 (Week 96) | 37.0 (3.13) | 11.4 (2.85)
  Anti-HPV-18 (Week 15): number analyzed (Participants) | 23 | 8
  Anti-HPV-18 (Week 15) | 24.8 (3.73) | 133.7 (4.32)
  Anti-HPV-18 (Week 27) | 44.7 (3.67) | 89.4 (4.85)
  Anti-HPV-18 (Week 48): number analyzed (Participants) | 20 | 8
  Anti-HPV-18 (Week 48) | 69.3 (3.87) | 133.7 (4.36)
  Anti-HPV-18 (Week 74): number analyzed (Participants) | 15 | 6
  Anti-HPV-18 (Week 74) | 83.2 (3.98) | 45.0 (4.23)
  Anti-HPV-18 (Week 96): number analyzed (Participants) | 3 | 4
  Anti-HPV-18 (Week 96) | 2.9 (1.86) | 2.2 (1.61)

12. Secondary Outcome: Change From Baseline in Flow Cytometry Response Magnitude
Description: Assessment of cellular immune activity was measured using the application of flow cytometry for the purpose of performing a Lytic Granule Loading Assay. The Lytic Granule Loading Assay examines the following external cellular markers: cluster of differentiation 3 (CD3), CD4, CD8 (T-cell identification), CD137, CD38, and CD69 (T-cell activation markers) as well as PD-1 (exhaustion/activation marker). Here, a change from baseline in CD8+/CD137+ PBMCs expressing Perforin+ was reported.
Time Frame: Baseline; Week 27
Population: as for outcome 1
Measure: Median (Full Range); unit: SFU/10^6 PBMC
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
Number analyzed (Participants) | 22 | 7
SFU/10^6 PBMC
  Baseline | 0.150 [0.00 to 14.50] | 1.250 [0.00 to 3.35]
  Change from Baseline at Week 27 | 0.000 [0.00 to 18.70] | 0.000 [0.00 to 7.70]

ADVERSE EVENTS:
Time Frame: From the first injection up to Week 100
Description: Safety population included all participants who received at least 1 dose of VGX-3100 (with or without EP).
Arm/Group | VGX-3100 + EP | VGX-3100 + EP + Imiquimod
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/25 | 0/8
Other Adverse Events (participants affected / at risk) | 23/25 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 + EP (N=25) | VGX-3100 + EP + Imiquimod (N=8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 + EP (N=25) | VGX-3100 + EP + Imiquimod (N=8)
Palpitations (Cardiac disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1
Vision blurred (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Injection site pain (General disorders) | 18 | 6
Fatigue (General disorders) | 14 | 4
Injection site swelling (General disorders) | 9 | 3
Injection site erythema (General disorders) | 8 | 3
Injection site bruising (General disorders) | 10 | 0
Injection site pruritis (General disorders) | 5 | 0
Malaise (General disorders) | 4 | 0
Pyrexia (General disorders) | 1 | 2
Influenza like illness (General disorders) | 0 | 2
Application site pain (General disorders) | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (General disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 1
Body temperature increased (Investigations) | 3 | 0
Weight increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 10 | 3
Dizziness (Nervous system disorders) | 4 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Vulvovaginal pruritis (Reproductive system and breast disorders) | 5 | 2
Vulvovaginal discomfort (Reproductive system and breast disorders) | 3 | 1
Vulval disorder (Reproductive system and breast disorders) | 3 | 0
Dyspareunia (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 2
Hot flush (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03180684/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT03180684/SAP_001.pdf